CLINICAL TRIAL: NCT00947934
Title: Study of the Effect of the Chronic Electric Stimulation of the Hypothalamus/Fornix on Memory Impairment in Alzheimer Disease.
Brief Title: Study of the Brain Stimulation Effect on Memory Impairment in Alzheimer Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: probleme of feasibility
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09 - APN - 04; AFSSAPS2009-A00318-49
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2009-07

CONDITIONS: Memory Disorders
Keywords: Alzheimer disease,hypothalamus,Deep Brain Stimulation
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep brain stimulation (Experimental): Electrodes (Medtronic 3389) will be implanted in a bilateral way , under local anesthesia, at fornix level in its way through the hypothalamus, very visible on the MRI just before its entrance to mammilary bodies. Electrodes will be connected under general anesthesia to the pectoral sub-cutaneous pacemaker. The electric chronic stimulation (180 Hz, 2-3 V, 120 ms) will be begun the day after the operation.
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Electrodes (Medtronic 3389) will be implanted in a bilateral way , under local anesthesia, at fornix level in its way through the hypothalamus, very visible on the MRI just before its entrance to mammilary bodies. Electrodes will be connected under general anesthesia to the pectoral sub-cutaneous pacemaker. The electric chronic stimulation (180 Hz, 2-3 V, 120 ms) will be begun the day after the operation
  Other Names: Hypothalamus/fornix stimulation; Medtronic 3389

SUMMARY:
Alzheimer's Disease (AD) is the most common cause of dementia. Today no treatment had shown consistent efficacy to stop or slow down the disease. Recent report of enhancement of memory abilities by bilateral chronic deep brain stimulation (DBS) of the fornix in the hypothalamus suggests that neuromodulation of circuits involved in memory processes may have therapeutic implications in AD patients with memory decline.

The primary objectives of this prospective, non-controlled, pilot study are to assess the feasibility and safety of DBS in AD patients with mild cognitive and memory impairment, and to evaluate the efficacy of DBS to slow down or stabilize this decline. Five patients with AD (DSM IV) diagnosed less than two years, with mild cognitive decline (MMSE 20-24), and specific impairment of episodic memory will be included in a 2-year period. The evaluation criteria for feasibility will be the proportion of patients undergoing the procedure, chronic stimulation and evaluation process without adverse event (AE). Efficacy will be evaluated using numerous cognitive and memory testing including classical instrument used in AD clinical trials. Changes in behavioral scales, and changes in hypothalamic functions (clinical, biological and hormonal assessment) will evaluate safety and tolerance. Clinical, neuro-psychological, biological and imaging assessment will be performed 3 and one month before and 3, 6, 12 and 24 months after surgery. Bilateral electrodes (Medtronic 3389) will be implanted, by MR-guided frame-based stereotaxy, in the hypothalamic part of the fornix, and then connected to the generator (Kinetra, Medtronic). Chronic high-frequency stimulation will be delivered immediately after surgery.

The investigators expect to slow down, or to stabilize the spontaneous decline of MMSE and ADAS scores after 6, 12 and 24 months of stimulation. In case of efficacy, DBS might offer to AD patient the possibility to slow down/stabilize their symptoms, which no other treatment can currently offer, and to increase their quality of life.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is the most common cause of dementia whom estimated prevalence rise to more than 5 millions in the US. AD patients display progressive impairment of episodic memory and instrumental signs including aphasia, apraxia, and agnosia, together with general cognitive decline, death occurring 6-9 years after diagnosis. Up to now, no treatment had shown consistent efficacy to stop or slow down the disease. Recently, it has been shown that memory abilities have been enhanced by bilateral chronic deep brain stimulation (DBS) of the fornix in the hypothalamus, in a patient initially treated for malignant obesity (Hamani C, Ann Neurol, 2008). This report showed that neuro-anatomic circuits involved in memory processes are reachable and can be modulated. This modulation may have therapeutic implications in AD patients with memory decline.

The primary objectives of this prospective, non-controlled, pilot study are to evaluate the feasibility and safety of DBS in AD patients with mild cognitive and memory impairment, and to evaluate the efficacy of DBS to slow down or stabilize this decline. The secondary objectives are to determine which cognitive and memory aspects are improved, and the duration of the efficacy of DBS on AD symptoms.

The inclusion criteria are: patients with AD (DSM IV) diagnosed less than two years, age between 50 and 65, with mild cognitive decline (MMSE between 20 and 24), and specific impairment of episodic memory (using the free and cued selective reminding test: FCSRT ), able to give and sign an informed consent. Patients with associated DSM I axis pathology, contra-indication to surgery or MRI, or preoperative MRI abnormalities will not be included. Five patients will be included in a 2-year period.

The evaluation criteria for feasibility will be the proportion of patients undergoing the procedure, chronic stimulation and evaluation process without adverse event (AE). Efficacy will be evaluated using numerous cognitive and memory testing including WAIS, MMSE, ADAS scales, TMT-A and TMT-B testing, language evaluation, FCSRT and Rey figure. CGI and IADL will evaluate global improvement. Neuro-imaging changes after stimulation will be evaluate by morphological MRI (hippocampal volume) and functional imaging (PET). Changes in behavioral and mood scales, and changes in hypothalamic functions (clinical, biological and hormonal assessment) will evaluate safety and tolerance.

Experimental paradigm: Clinical, neuro-psychological, biological and imaging assessment will be performed 3 and one month before and 3, 6, 12 and 24 months after surgery. Bilateral electrodes (Medtronic 3389) will be implanted, under local anesthesia, by MR-guided frame-based stereotaxy, in the hypothalamic part of the fornix, before its entry in the mamillary body (well defined on T2 weighted sequences). Intraoperative stimulation will be used to search adverse effects or acute effects. Electrodes will be connected to the generator (Kinetra, Medtronic) under general anesthesia. Chronic high-frequency stimulation will be delivered immediately after surgery.

Expected results and perspectives: Spontaneously, neuropsychological scores progressively decline with time in AD patients (MMSE 3-4 points decrease and ADAS 6 points increase per year). We expect to slow down, or to stabilize these scores after 6, 12 and 24 months of stimulation.

In case of efficacy DBS might offer to AD patient the possibility to slow down/stabilize their symptoms, which no other treatment can currently offer, and to increase their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 50 and 65 years of age,
* Patients with Alzheimer disease (according to DSM-IV criteria)
* Recent diagnosis of Alzheimer disease (less than 2 years ago)
* Patients with a total score in "Mini Mental Test" between 20 and 24.
* Patient with impaired performance of their occasional memory, estimated by the test of Grober and Buschke (according to the standards, according to the age, the sex and the sociocultural level).
* Patients covered by Social Security
* Patients willing to sign the proper consent forms

Exclusion Criteria:

* associated DSM I axis pathology,
* contra-indication to surgery or MRI,
* preoperative MRI abnormalities
* Withdrawal of patient consent
* Study sponsor or investigator decision to suspend the study.
* Diagnosis of a metabolic or hormonal disorder on the biological assessment realized during the inclusion.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Evaluation criteria for feasibility will be the proportion of patients undergoing the procedure, chronic stimulation and evaluation process without adverse event. | 2012

SECONDARY OUTCOMES:
- Efficacy : evaluated using cognitive and memory testing. - Global improvement : CGI and IADL - Neuro-imaging : MRI and functional imaging - Safety/tolerance : Changes in behavioral,in hypothalamic functions and assessment of adverse events | 2012

CONTACTS AND LOCATIONS:
Overall Officials: Denys Fontaine, PH, Principal Investigator — Service de Neurochirurgie; Philippe Robert, PH PU, Principal Investigator — CMR2
Locations (2):
- France (2):
  - CMR2 Hôpital de Cimiez, Nice
  - Service de Neurochirurgie Hôpital Universitaire de Pasteur, Nice